CLINICAL TRIAL: NCT00708344
Title: Efficacy and Safety of Irbesartan/Hydrochlorothiazide Combination: A Comparison of Active and Usual Titration Regimen in the Treatment of Hypertensive Patients Insufficiently Controlled by Monotherapy
Brief Title: ACTUAL: Efficacy and Safety of Irbesartan/Hydrochlorothiazide Combination
Acronym: ACTUAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBEH_R_02931
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Usual elective titration regimen
  Interventions: Drug: Irbesartan - Hydrochlorothiazide
- Group 2 (Active Comparator): Active elective titration regimen
  Interventions: Drug: Irbesartan - Hydrochlorothiazide

INTERVENTIONS:
Drug: Irbesartan - Hydrochlorothiazide — 150/12.5 mg (1 tablet once daily) or 300/25 mg (1 tablet once daily) depending on the control of the blood pressure. Duration of treatment : 10 weeks
  Arms: Group 1
Drug: Irbesartan - Hydrochlorothiazide — 150/12.5 mg (1 tablet once daily) or 300/25 mg (1 tablet once daily) depending on the control of the blood pressure. Treatment duration : 10 weeks
  Arms: Group 2

SUMMARY:
To compare the antihypertensive efficacy of the combination irbesartan/hydrochlorothiazide (HCTZ) using either a usual or an active elective titration regimen. The main efficacy criteria will be the change in mean Systolic Blood Pressure (SBP), measured at doctor's office with an automatic device, after a 10-week treatment period in hypertensive patients insufficiently controlled by monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Established essential hypertension treated for at least 4 weeks by one antihypertensive drug alone
* With uncontrolled Blood Pressure (BP) defined as:
* SBP ≥ 160 mmHg and/or DBP ≥ 100 mmHg in non diabetic patients
* SBP ≥ 150 mmHg and/or DBP ≥ 90 mmHg in diabetic patients

Exclusion Criteria:

* SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg at V1
* Known or suspected causes of secondary hypertension
* Patient with bilateral renal artery stenosis, renal artery stenosis in a solitary kidney; history of renal transplant or only has one functioning kidney
* Associated cardiovascular conditions that prevent the patient from stopping the current antihypertensive drug (e.g.: Beta-blocker for angina, ACE-inhibitors for heart failure, etc…).
* Known hypersensitivity to diuretics or sulphonamides or history of angioedema or cough related to the administration of an angiotensin II receptor antagonist or any combination of the drugs used
* Known contraindications to the study drugs:
* Severe renal dysfunction (creatinine clearance <30ml/min)
* Known hypokaliemia (< 3 mmol/L) , known hypercalcemia
* Severe hepatic impairment, biliary cirrhosis, cholestasis
* Inability to obtain a valid automatic BP measurement recording
* Administration of any other investigational drug within 30 days prior to study entry and during the course of the study
* Presence of any severe medical or psychological condition that, in the opinion of the investigator, indicate that participation in the study is not in the best interest of the subject.
* Presence of any other conditions (e.g. geographic, social, etc) that would restrict or limit the subject participation for the duration of the study.
* Pregnant or breast-feeding women
* Women of childbearing potential not protected by effective contraceptive method of birth control

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Change in mean Systolic Blood Pressure | between Visit 1 (Week 0) and Visit 4 (Week 10)

SECONDARY OUTCOMES:
Change in mean Diastolic Blood Pressure | between Visit 1 (Week 0) and Visit 4 (Week 10)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie - GENES, MD, Study Director — Sanofi
Locations (16):
- Sanofi-Aventis Administrative Office, Algiers, Algeria
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Quito, Ecuador
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Guatemala City, Guatemala
- Sanofi-Aventis Administrative Office, Beirut, Lebanon
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico
- Sanofi-Aventis Administrative Office, Casablanca, Morocco
- Sanofi-Aventis Administrative Office, Panama City, Panama
- Sanofi-Aventis Administrative Office, Lima, Peru
- Sanofi-Aventis Administrative Office, Jeddah, Saudi Arabia
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Dubai, United Arab Emirates
- Sanofi-Aventis Administrative Office, Caracas, Venezuela

REFERENCES:
- [Derived] Girerd X, Rosenbaum D, Aoun J; ACTUAL study Investigators. Efficacy and safety of early versus late titration of fixed-dose irbesartan/hydrochlorothiazide: ACTUAL study. Blood Press Suppl. 2011 Dec;2:22-9. doi: 10.3109/08037051.2011.633368. PMID 22352122